CLINICAL TRIAL: NCT04650581
Title: Double-Blind Placebo-Controlled Randomized Phase III Trial of Fulvestrant and Ipatasertib as Treatment for Advanced HER-2 Negative and Estrogen Receptor Positive (ER+) Breast Cancer Following Progression on First Line CDK 4/6 Inhibitor and Aromatase Inhibitor
Brief Title: Fulvestrant and Ipatasertib for Advanced HER-2 Negative and Estrogen Receptor Positive (ER+) Breast Cancer Following Progression on First Line CDK 4/6 Inhibitor and Aromatase Inhibitor
Acronym: FINER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA40; 2101 (Other: BCT); M041883 (Other: Hoffmann-LaRoche Ltd.)
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipatasertib + Fulvestrant (Experimental)
  Interventions: Drug: Ipatasertib; Drug: Fulvestrant
- Placebo (Placebo Comparator)
  Interventions: Drug: Fulvestrant; Other: Placebo

INTERVENTIONS:
Drug: Ipatasertib — 400 mg PO QD days 1-21 every 28 days
  Arms: Ipatasertib + Fulvestrant
Drug: Fulvestrant — 500 mg IM cycle 1 days 1 and 15 followed by 500 mg IM day 1 q 28 days subsequent cycles
Other: Placebo — PO QD days 1-21 every 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether a new drug, Ipatasertib, can slow the growth of advanced breast cancer when added to standard therapy (Fulvestrant).

DETAILED DESCRIPTION:
Patients enrolled in this study will receive either Ipatasertib plus Fulvestrant or placebo (a substance that looks like the study drug but does not have any active or medicinal ingredient) plus Fulvestant. The study will provide information about the ability of Ipatasertib plus Fulvestrant to control the cancer, the side effects and safety of the treatment, how patients feel while taking the treatment and associated costs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed ER positive, HER-2 negative breast cancer
* Female patients must be post-menopausal; female patients who are pre-menopausal must have ovarian suppression using LHRH agonist while on study
* Clinical and/or radiographic progression during treatment with or within 28 days after discontinuation of first line of treatment with a CDK 4/6 inhibitor and an aromatase inhibitor (AI) for advanced/metastatic disease
* Evidence of clinically and/or radiologically documented disease
* ≥ 18 years of age
* ECOG performance status of 0 or 1
* No concurrent anti-cancer therapy and must satisfy the following criteria for previous therapy

  * Must not have received more than one prior line of treatment with a CDK 4/6 inhibitor and an AI in the advanced disease setting.
  * Treatment with CDK 4/6 inhibitor and AI must have been the most recent treatment prior to registration for this study
* Adequate hematology and organ function, in the absence of growth factors

  * Absolute neutrophils > 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Hemoglobin > 90 g/L
  * Total Bilirubin ≤ 1.5 x ULN (upper limit of normal) or ≤ 3 x ULN if confirmed Gilbert's Syndrome
  * ALT and AST ≤ 2.5 x ULN (or ≤ 5.0 x ULN if liver or bone metastasis)
  * Alkaline phosphatase ≤ 2.0 x ULN (or ≤ 5.0 x ULN if liver metastases, ≤ 7.0 x ULN if bone metastasis)
  * Fasting glucose ≤ 8.3 mmol/L
  * HbA1c ≤ 7.5%
  * Serum albumin ≥ 30 g/L
  * INR ≤ 1.2
  * Serum Creatinine or Creatinine clearance ≤ 1.5 x ULN or ≥ 50 mL/min; measured directly by 24-hour urine sampling or as calculated by Crockcroft and Gault equation

Exclusion Criteria:

* Untreated or symptomatic CNS metastases, radiation treatment for CNS metastases within 28 days
* Active inflammatory bowel disease, bowel inflammation, inability to swallow oral medication or GI condition that alters oral absorption
* Prior treatment with fulvestrant, selective estrogen receptor degraders (SERDs) or known inhibitors of the PI3K pathway including PI3K inhibitors, AKT inhibitors, or mTOR inhibitors
* Mean QT interval corrected for heart rate (QTc) ≥ 480 msec by ECG or history of familial long QT syndrome
* Active or uncontrolled infections or serious illnesses or medical conditions
* Clinically significant liver diseases
* History of lung disease or history of opportunistic infections
* Type 1 or Type 2 diabetes mellitus requiring insulin
* Grade ≥ 2 uncontrolled hypercholesterolemia or hypertriglyceridemia
* Known abnormalities in coagulation
* History of hypersensitivity to the study drugs or components
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chia, Study Chair — BCCA - Vancouver Cancer Centre, BC Canada
Locations (39):
- Australia (16):
  - Southern Highlands Cancer Centre, Bowral, New South Wales
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Macquarie University Hospital, Macquarie University, New South Wales
  - Shoalhaven Cancer Care Centre, Nowra, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Victorian Breast and Oncology Care, East Melbourne, Victoria
  - The Northern Hospital, Epping, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - St John of God Bunbury, Bunbury, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Canberra Hospital, Garran
  - Royal Brisbane and Womens Hospital, Herston
- Canada (21):
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health System, Brampton, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Sciences Centre/, Thunder Bay, Ontario
  - University Health Network, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Centre Integre de Sante et de Services Sociaux, Greenfield Park, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Wellington Cancer Centre, Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: January 27, 2021 to May 08, 2024
Groups:
- Ipatasertib + Fulvestrant: Ipatasertib will be administered orally at a dose of 400 mg once daily from Day 1 to Day 21 of each cycle. Fulvestrant will be administered intramuscularly at a dose of 500 mg. For the first cycle only, fulvestrant will be given on both Day 1 and Day 15. In all subsequent cycles, fulvestrant will be administered on Day 1 only. The duration of each cycle is 28 days.
- Placebo + Flvestrant: Placebo will be administered orally at a dose of 400 mg once daily from Day 1 to Day 21 of each cycle. Fulvestrant will be administered intramuscularly at a dose of 500 mg. For the first cycle only, fulvestrant will be given on both Day 1 and Day 15. In all subsequent cycles, fulvestrant will be administered on Day 1 only. The duration of each cycle is 28 days.
Period: Overall Study
Arm/Group | Ipatasertib + Fulvestrant | Placebo + Flvestrant
Started | 125 | 125
Completed | 124 | 124
Not Completed | 1 | 1
Not completed — No treated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipatasertib + Fulvestrant | Placebo + Flvestrant | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Continuous [Median (Full Range); unit: Years] — Age measured in years
  Years | 60 [29 to 89] | 59 [33 to 83] | 60 [29 to 89]
Sex: Female, Male [Count of Participants; unit: Participants] — Biological Sex such as female and male
  Participants
    Female | 123 | 124 | 247
    Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race defined by the national institutes of health
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 16 | 12 | 28
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 4 | 1 | 5
    White | 98 | 107 | 205
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: Participants] — Country or region of enrollment
  Participants
    Canada | 89 | 91 | 180
    Australia | 29 | 29 | 58
    New Zealand | 7 | 5 | 12
Body Mass Index [Mean (Standard Deviation); unit: Kg per meter square (kg/(m*m))] — BMI (Body Mass Index) is a measurement that helps determine if a person has a healthy weight for their height. It is calculated by dividing a person's weight in kilograms by their height in meters squared. Population: Intent to treat
  Kg per meter square (kg/(m*m)) | 27.72 (5.68) | 27.26 (5.29) | 27.49 (5.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival (PFS) Using RECIST 1.1
Description: Progression-free survival (PFS) defined as time from randomization to disease progression or death from any cause, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 4 years
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Ipatasertib + Fulvestrant | Placebo + Flvestrant
Number analyzed (Participants) | 125 | 125
Participants | 94 | 103
Statistical Analysis 1: Comparison: Ipatasertib + Fulvestrant vs Placebo + Flvestrant; Test type: Superiority; p = 0.0007, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.46 to 0.81]

2. Secondary Outcome: To Compare the Two Treatment Arms With Respect to Investigator Assessed PFS (Per RECIST 1.1) in the PIK3CA/AKT1/PTEN Altered Cohort
Description: The PFS is tested in the PIK3CA/PTEN/AKT1 altered status subset under the same 0.05 significance level among the 111 subjects in the PIK3CA/PTEN/AKT1 altered status subset
Time Frame: 4 years
Population: Subset of patients in the PIK3CA/AKT1/PTEN altered cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Ipatasertib + Fulvestrant | Placebo + Flvestrant
Number analyzed (Participants) | 57 | 54
Participants | 43 | 50
Statistical Analysis 1: Comparison: Ipatasertib + Fulvestrant vs Placebo + Flvestrant; Test type: Superiority; p = 0.0005, Log Rank; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.31 to 0.72]

3. Secondary Outcome: Commencement of Subsequent Line of Systemic Therapy or Death (TSST)
Description: Number of patients with commencement of subsequent line of systemic therapy or death between enrollment and the end of study
Time Frame: 4 years
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Ipatasertib + Fulvestrant | Placebo + Flvestrant
Number analyzed (Participants) | 125 | 125
Participants | 95 | 98
Statistical Analysis 1: Comparison: Ipatasertib + Fulvestrant vs Placebo + Flvestrant; Test type: Superiority; p = 0.0075, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.51 to 0.90]

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 4 years
Description: All-cause mortality was analyzed based on all 250 randomized patients. Serious Adverse Events and Other Adverse Events were analyzed based on 248 patients who received protocol treatment.
Arm/Group | Ipatasertib + Fulvestrant | Placebo + Flvestrant
All-Cause Mortality (participants affected / at risk) | 42/125 | 36/125
Serious Adverse Events (participants affected / at risk) | 18/124 | 18/124
Other Adverse Events (participants affected / at risk) | 124/124 | 120/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipatasertib + Fulvestrant (N=124) | Placebo + Flvestrant (N=124)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Death NOS (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Uterine perforation (Injury, poisoning and procedural complications) | 5 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipatasertib + Fulvestrant (N=124) | Placebo + Flvestrant (N=124)
Palpitations (Cardiac disorders) | 3 | 7
Abdominal pain (Gastrointestinal disorders) | 30 | 21
Bloating (Gastrointestinal disorders) | 15 | 16
Constipation (Gastrointestinal disorders) | 45 | 61
Diarrhea (Gastrointestinal disorders) | 112 | 44
Dry mouth (Gastrointestinal disorders) | 14 | 10
Dyspepsia (Gastrointestinal disorders) | 7 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 11 | 13
Mucositis oral (Gastrointestinal disorders) | 25 | 11
Nausea (Gastrointestinal disorders) | 96 | 57
Vomiting (Gastrointestinal disorders) | 56 | 26
Edema limbs (General disorders) | 11 | 12
Fatigue (General disorders) | 83 | 77
Fever (General disorders) | 10 | 11
Flu like symptoms (General disorders) | 6 | 7
Injection site reaction (General disorders) | 4 | 12
Non-cardiac chest pain (General disorders) | 10 | 11
Pain (General disorders) | 23 | 20
Other infections and infestations (Infections and infestations) | 15 | 12
Upper respiratory infection (Infections and infestations) | 9 | 8
Urinary tract infection (Infections and infestations) | 9 | 7
Anorexia (Metabolism and nutrition disorders) | 38 | 24
Dehydration (Metabolism and nutrition disorders) | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 49
Bone pain (Musculoskeletal and connective tissue disorders) | 45 | 43
Buttock pain (Musculoskeletal and connective tissue disorders) | 9 | 10
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 31
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 24
Dizziness (Nervous system disorders) | 18 | 17
Dysgeusia (Nervous system disorders) | 13 | 6
Headache (Nervous system disorders) | 48 | 41
Neuralgia (Nervous system disorders) | 7 | 5
Paresthesia (Nervous system disorders) | 10 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 19
Anxiety (Psychiatric disorders) | 22 | 17
Depression (Psychiatric disorders) | 5 | 7
Insomnia (Psychiatric disorders) | 35 | 36
Breast pain (Reproductive system and breast disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 22
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 35 | 36
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 13
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 12
Rash acneiform (Skin and subcutaneous tissue disorders) | 13 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 35 | 15
Hot flashes (Vascular disorders) | 25 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT04650581/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT04650581/SAP_001.pdf